CLINICAL TRIAL: NCT01034371
Title: Comparison of "One-stop" Hybrid Coronary Revascularization Versus Off-pump Coronary Artery Bypass for the Treatment of Multi-vessel Coronary Artery Disease
Brief Title: Comparison of One-stop Hybrid Revascularization Versus Off-pump Coronary Artery Bypass for the Treatment of Multi-vessel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: China National Center for Cardiovascular Diseases ( Shengshou Hu MD, FACC ), China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20091216
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2009-12-21 (Estimated); Status verified 2009-12

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Hybrid Revascularization;; Percutaneous Coronary Intervention; Coronary Artery Bypass
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Artery Bypass, Off-Pump

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- One-stop hybrid revasularization (Experimental)
  Interventions: Procedure: Minimally invasive direct coronary artery bypass; Procedure: PCI-Drug eluting stents
- Off-pump coronary artery bypass (Active Comparator)
  Interventions: Procedure: Off-pump coronary artery bypass

INTERVENTIONS:
Procedure: Minimally invasive direct coronary artery bypass — MIDCAB with no associated or concomitant surgical procedures, using partial ministernotomy, without cardiopulmonary bypass (CPB) and cardioplegia.
  Other Names: MIDCAB
  Arms: One-stop hybrid revasularization
Procedure: PCI-Drug eluting stents — PCI with drug eluting stents (DES) performed by cardiologists on the non-LAD lesions in the same operating suite immediately following MIDCAB.
  Device: Polymer-based Sirolimus-Eluting Stents (SES).
  Other Names: PCI
  Arms: One-stop hybrid revasularization
Procedure: Off-pump coronary artery bypass — Procedure: coronary artery bypass without cardiopulmonary Coronary artery bypass surgery with no associated or concomitant surgical procedures, using full median sternotomy, without cardiopulmonary bypass (CPB) and cardioplegia.
  Other Names: OPCAB
  Arms: Off-pump coronary artery bypass

SUMMARY:
The "one-stop" hybrid coronary revascularization combines minimally invasive direct coronary artery bypass (MIDCAB) and PCI to be performed in the hybrid operating suite, an enhanced operating room equipped with radiographic capability. This study is to compare 1-year clinical outcomes of "one-stop" hybrid coronary revascularization with off-pump coronary artery bypass (OPCAB) in selected patients with multivessel coronary artery disease.

DETAILED DESCRIPTION:
- With the development of specialized devices and experience, off-pump coronary artery bypass (OPCAB) has been a well-established less invasive technique for coronary revascularization. Compared with conventional on-pump coronary artery bypass grafting (CABG), OPCAB avoids the use of cardiopulmonary bypass and cardioplegic arrest, and is associated with decreased morbidity, shorter length of stay in ICU and hospital, and less perioperative complications, especially in elderly patients with severe comorbidities. "One-stop" (also named simultaneous) hybrid coronary revascularization is also a novel, safe and feasible minimally invasive approach in selected patients with multivessel coronary artery disease (CAD). It allows surgical and interventional procedures to be performed consecutively in the "one-stop" hybrid operating suite, an enhanced operating room equipped with radiographic capability, wherein the left intramammary artery (LIMA) is placed on the left anterior descending artery (LAD) by minimally invasive procedure, immediately followed by percutaneous coronary intervention/stenting on the non-LAD lesions. However, few studies are now available on the outcomes of coronary revascularization between the new hybrid strategy with conventional OPCAB. This study is a single center randomized clinical trial to compare 1-year clinical outcomes of "one-stop" hybrid coronary revascularization with OPCAB in selected patients with multivessel CAD with suitable coronary anatomy.

Sample size:

- We examined the results of SYNTAX trial and of our institution published previously. The 1-year MACCE rate (the primary endpoint) is estimated as being 13% for OPCAB. The sample calculated for this trial is 400 patients.

Design/Methodology:

- Trial design: A single center randomized clinical trial comparing "one-stop" hybrid procedure versus conventional OPCAB in 400 patients with suitable anatomy who need revascularization.

Intervention: Patients will be randomized to undergo either "one-stop" hybrid procedure or conventional OPCAB.

- Randomization: Patients will be evaluated by both a cardiac surgeon and an interventional cardiologist. After obtaining informed written consent, patients will be randomized to receive "one-stop" hybrid procedure or conventional OPCAB. An expertise-based randomization will be used.

The data adjudicators will be blinded to the study. Due to the nature of this study, the operating surgeons, cardiologists, anesthetists, other operative room staff, and ICU staff will not be blind in this study.

Study intervention:

- Candidates will be randomized to receive "one-stop" hybrid procedure or conventional OPCAB.

ELIGIBILITY:
Inclusion Criteria:

* Two- or three-vessel disease, left main disease, or LM equivalent with 2 or 3-vessel disease (left anterior descending [LAD], left circumflex [LCX], right coronary artery [RCA] territory);
* LAD diseases not suitable for PCI [i.e. chronic totally occlusion (CTO), severe calcification or/and angulated lesions, bifurcation or trifurcation lesions];
* Angiographic characteristics of non-LAD lesion(s) amiable to PCI;
* Chronic stable or unstable angina pectoris of CCS 2 or greater (symptoms of angina and/or objective evidence of myocardial ischemia);
* Evaluated by both cardiac surgeon and cardiologist together.

Exclusion Criteria:

* Need for emergent CABG;
* Prior CABG;
* Prior PCI with stenting within 6 months of study entry;
* Stroke with 6 months of study entry;
* Overt congestive heart failure;
* Need for a concomitant operation (i.e. valve repair or replacement, Maze surgery);
* Hemodynamic instability;
* Situations in which complete revascularization is not possible served;
* Allergy to radiographic contrast, aspirin or clopidogrel.
* Contradictions to PCI: Occluded coronary vessels, PVD, Unable to achieve access, Fresh thrombus, Vessels <1.5mm; Intolerance to aspirin or both clopidogrel and ticlopidine;
* Cannot undergo either CABG or PCI/DES because of a coexisting medical condition
* History of significant bleeding; Significant leukopenia, neutropenia, thrombocytopenia, anemia, or known bleeding diathesis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2009-12; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Composite of major adverse cardiac or cerebrovascular events (MACCE) including death, myocardial infarction, stroke and/or repeat revascularization. | 1 year

SECONDARY OUTCOMES:
Overall MACCE rate. | 30 days after procedure and 2 years after enrollment
Cardiac death. | 30 days after procedure, 1 and 2 years after enrollment
Documented myocardial infarction. | 30 days after procedure, 1 and 2 years after enrollment
Target lesion revascularization. | 30 days after procedure, 1 and 2 years after enrollment
Recurrence of Angina. | 1 and 2 years after enrollment
Cost-effectiveness analysis. | 1 and 2 years after enrollment
Quality of life. | 6 months, 1 and 2 years after enrollment
Rehospitalization. | 6 months, 1 and 2 years after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Shengshou Hu, M.D., Study Director — China National Center for Cardiovascular Diseases
Locations (2):
- China (2):
  - China National Center for Cardiovascular Diseases, Cardiovascular Institute & Fuwai Hospital, Beijing, Beijing Municipality
  - Institute of cardiovascular diseases & Fuwai hospital, Beijing, Beijing Municipality